CLINICAL TRIAL: NCT06709534
Title: Feasibility and Acceptability of an Individualized Online Home-Based Exercise Program on Psychoneurological Symptoms in Gynecologic Cancer Survivors: A Pilot Study
Brief Title: An Individualized Online Home-Based Exercise Program for Improving Symptoms in Gynecologic Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Zahra A. Barandouzi, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00007783; P30CA138292 (NIH); NCI-2024-08387 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EU6320-24 (Other: Emory University Hospital/Winship Cancer Institute)
Record Dates: First submitted 2024-10-25; First posted 2024-11-29 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Malignant Female Reproductive System Neoplasm
MeSH Terms: interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (individualized online home-based exercise) (Experimental): Participants meet with a certified exercise trainer and complete a functional capacity assessment using a treadmill or 6-minute walk test. Participants then complete an individualized online home-based exercise intervention via Zoom consisting of progressive, moderate-intensity walking corresponding to the RPE scale and receive social support over 30 minutes BIW for 12 weeks.
  Interventions: Other: Exercise Intervention; Other: Functional Assessment; Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration; Other: Supportive Care

INTERVENTIONS:
Other: Exercise Intervention — Participate in an individualized online home-based exercise intervention
Other: Functional Assessment — Complete functional capacity assessment
Other: Medical Device Usage and Evaluation — Wear an activity tracker
Other: Questionnaire Administration — Ancillary studies
Other: Supportive Care — Receive social support
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive

SUMMARY:
This clinical trial tests an individualized online home-based exercise program in gynecologic cancer survivors and its impact on gut microbiome (the bacteria and microorganisms that live in the digestive system) and symptoms such as pain, fatigue, sleep disturbance, depression, and cognitive impairment. These symptoms can significantly reduce the quality of life (QoL) and survival rate in this cancer population. Thus, promoting physical activity among cancer survivors may help mitigate these severe symptoms. Using online platforms such as Zoom can help participants access an individualized exercise program that meets their specific needs to engage in physical activity and decrease their symptom burden. Home-based exercise, by providing self-chosen time and location and low costs, can address some barriers to physical activity for cancer survivors. An individualized online home-based exercise program may be feasible, and may improve symptoms and quality of life in gynecologic cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine the feasibility and acceptability of an individualized home-based exercise program in gynecologic cancer survivors.

II. To test the effect of the program on gut microbiome and psychoneurological symptoms in gynecologic cancer survivors.

OUTLINE:

Participants meet with a certified exercise trainer and complete a functional capacity assessment using a treadmill or 6-minute walk test. Participants then complete an individualized online home-based exercise intervention via Zoom consisting of progressive, moderate-intensity walking corresponding to the rate of perceived exertion (RPE) scale and receive social support over 30 minutes twice a week (BIW) for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 years old
* Previously diagnosed with gynecologic cancer (e.g., uterine, ovarian, cervical)
* Completed cancer treatment (chemotherapy or chemoradiation)
* Able to read and speak English
* Do not meet recommended exercise levels as defined by The American College of Sports Medicine

Exclusion Criteria:

* History of metastatic or other primary cancer
* Serious mental health conditions (e.g., bipolar disorder, schizophrenia, major depression)
* Certain chronic diseases (e.g., muscular-skeletal diseases that limit mobility, autoimmune diseases, uncontrolled diabetes, hypertension, renal disease (creatinine > 2.5 mg/dL)
* Unable to read/speak English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Attrition Rates (Feasibility) | At 12 weeks
  Feasibility will be assessed by calculating attrition and adherence rates, identifying reasons for refusal, and evaluating the completeness of the data. We will consider the intervention to have low attrition and high adherence if >80% of participants remain enrolled and complete the study, respectively.
Adherence Rates (Feasibility) | At 12 weeks
  Feasibility will be assessed by calculating attrition and adherence rates, identifying reasons for refusal, and evaluating the completeness of the data. We will consider the intervention to have low attrition and high adherence if > 80% of participants remain enrolled and complete the study, respectively.
Intervention Acceptability | Up to 12 weeks
  Will be evaluated with a survey to assess participants' perceptions of the acceptability of the study procedures. A response rate of > 80% will be considered high acceptability. Descriptive statistics will be calculated using SPSS and R software.
Gut Microbiome | From baseline to 12 weeks
  Gut microbiota composition will be evaluated using collected stool samples. The preliminary efficacy of the intervention on gut microbiome and psychoneurological symptoms (PNS) will be compared using a paired t-test.
Psychoneurological Symptoms | From baseline to 12 weeks
  Will be assessed using the Fatigue Short Form, Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress-Depression and Anxiety Short Form, Pain Interference Short Form, PROMIS Cognitive Function Short Form, PROMIS Sleep Disturbance Short Form, the PROMIS gastrointestinal (GI) constipation and diarrhea Short Forms. The preliminary efficacy of the intervention on gut microbiome and PNS will be compared using a paired t-test.

SECONDARY OUTCOMES:
Quality of Life Assessment | Up to 12 weeks
  Quality of life will be assessed using the Short Form-8 questionnaire. The preliminary efficacy of the intervention on quality life will be compared using a paired t-test.
Rapid Eating Assessment for Participants | Up to 12 weeks
  Rapid Eating Assessment for Participants will be used to evaluate their diet. Diet will be assessed to control this variable for measuring gut microbiome.
Stress | Up to 12 weeks
  Stress level will be measured using PSS. The preliminary efficacy of the intervention on stress will be compared using a paired t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Zahra A Barandouzi, Ph.D.,MSN,RN, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (4):
- United States (4):
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Decatur Hospital, Decatur, Georgia